CLINICAL TRIAL: NCT00567671
Title: Safety and Effectiveness of the UV-X System for Corneal Collagen Cross-Linking in Eyes With Corneal Ectasia or Progressive Keratoconus
Brief Title: Corneal Collagen Cross-Linking for the Treatment of Progressive Keratoconus and Corneal Ectasia
Acronym: CL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: R. Doyle Stulting, MD, PhD., Professor of Ophthalmology, Emeritus, Principle Investigator, Woolfson Eye Intitute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UVX-001
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2009-07

CONDITIONS: Progressive Keratoconus; Corneal Ectasia
Keywords: keratoconus; ectasia; cross-linking; riboflavin; UVA light; cornea
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic; Corneal Diseases | interventions — Corneal Cross-Linking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Corneal collagen cross-linking
  Interventions: Procedure: Corneal collagen
- Control (Sham Comparator): Sham Treatment
  Interventions: Procedure: Sham comparator

INTERVENTIONS:
Procedure: Corneal collagen — Corneal collagen cross-linking with riboflavin/UVA light
  Arms: Treatment
Procedure: Sham comparator — Sham treatment
  Arms: Control

SUMMARY:
Prospective, randomized, single site study to determine the safety and effectiveness of performing corneal collagen cross-linking (CCCL)using riboflavin and UVA light in eyes with corneal ectasia or progressive keratoconus.

DETAILED DESCRIPTION:
Subjects are randomized to a control group or a treatment group, with the control group crossed over to the treatment group at the 3 month visit. Corneal collagen cross-linking is performed as a single treatment. Subjects are followed for at least 12 months to evaluate the long term effects of corneal collagen cross-linking.

Subjects may be referred from other physicians but must return to Emory Vision for completion of all study visits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of keratoconus with documented progression over the previous 12 months.
* Diagnosis of corneal ectasia
* Must be able to complete all study visits

Exclusion Criteria:

* Prior corneal surgery in the keratoconus group
* Corneal scarring

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change in keratometry | 3 Months

SECONDARY OUTCOMES:
Best spectacle-corrected visual acuity | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: R. Doyle Stulting, MD, PhD, Principal Investigator — Emory Vision; Emory University
Locations (1):
- Woolfson Eye Institute, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Hallahan KM, Rocha K, Roy AS, Randleman JB, Stulting RD, Dupps WJ Jr. Effects of corneal cross-linking on ocular response analyzer waveform-derived variables in keratoconus and postrefractive surgery ectasia. Eye Contact Lens. 2014 Nov;40(6):339-44. doi: 10.1097/ICL.0000000000000090. PMID 25365551
- See also: Click here to contact the investigator site for this study. — http://www.emoryvision.com